CLINICAL TRIAL: NCT04502992
Title: Neural Mechanisms of Acceptance and Commitment Therapy for Chronic Pain: A Network-Based fMRI Approach
Brief Title: Acceptance and Commitment Therapy, a Mindfulness-Based Approach for Treatment of Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Semra Aytur, Associate Professor, University of New Hampshire
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UNH-06-6991-01
Record Dates: First submitted 2020-07-23; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Chronic Musculoskeletal Disease
Keywords: Acceptance and commitment therapy; chronic pain; brain networks; functional connectivity; graph theory; fMRI
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Pre-post (quasi-experimental) design assessing the neural mechanisms underlying and behavioral changes associated with a 4 week Acceptance and Committment Therapy (ACT) intervention among participants with chronic musculoskeletal pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (pre-post, quasi-experimental) (Other): Pre-post intervention, single arm. (Intervention was 4 weeks of Acceptance and Committment therapy, 2 times per week, 90 min per session, in a group setting).
  Interventions: Behavioral: Acceptance and Committment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Committment Therapy — Acceptance and Commitment Therapy (ACT) is a mindfulness-based therapy that focuses on enabling individuals to accept what is out of their control, and to commit to valued actions that enrich their lives (Vowles & McCracken, 2008). By emphasizing acceptance instead of avoidance, ACT differs from many other forms of cognitive behavioral therapy. ACT has been shown to be efficacious in terms of clinical outcomes, adherence to treatment, and retention. ACT aims to increase psychological flexibility, and has been associated with improved health outcomes prior randomized controlled clinical trials, including three systematic reviews specific to CP. Psychological flexibility is defined as an individual's ability to recognize and adapt to various demands; shift mindsets or behavioral responses when these strategies compromise personal or social functioning; and maintain balance among important life domains.

SUMMARY:
Acceptance and Commitment Therapy (ACT) has been recognized as an effective, non-pharmacologic treatment for a variety of CP conditions. However, little is known about the neurologic mechanisms underlying ACT. The investigators conducted an ACT intervention in women (n=9) with chronic musculoskeletal pain. Functional magnetic resonance imaging (fMRI) data were collected pre- and post-ACT, and changes in functional connectivity (FC) were measured using Network-Based Statistics (NBS). Behavioral outcomes were measured using validated assessments such as the Acceptance & Action Questionnaire (AAQ-II), the Chronic Pain Acceptance Questionnaire (CPAQ), the Center for Epidemiologic Studies Depression Scale (CES-D), and the NIH Toolbox Neuro-QoLTM (Quality of Life in Neurological Disorders) scales.

Results suggest that, following the four-week ACT intervention, participants exhibited reductions in brain activation within and between key networks including self-reflection (default mode, DMN), emotion (salience, SN), and cognitive control (frontal parietal, FPN). These changes in connectivity strength were correlated with changes in behavioral outcomes including decreased depression and pain interference, and increased participation in social roles. This study is one of the first to demonstrate that improved function across the DMN, SN, and FPN may drive the positive outcomes associated with ACT. This study contributes to the emerging evidence supporting the use of neurophysiological indices to characterize treatment effects of alternative and complementary mind-body therapies.

DETAILED DESCRIPTION:
Over 100 million Americans suffer from chronic pain (CP), which causes more disability than any other medical condition in the U.S. at a cost of $560-$635 billion per year. Opioid analgesics are frequently used to treat CP. However, long term use of opioids can cause brain changes such as opioid-induced hyperalgesia that, over time, increase pain sensation. Also, opioids fail to treat complex psychological factors that worsen pain-related disability, including beliefs and emotional responses to pain. Cognitive behavioral therapy (CBT) can be efficacious for CP. However, CBT does not focus on important factors needed for long-term functional improvement, including attainment of personal goals and the psychological flexibility to choose responses to pain.

Acceptance and Commitment Therapy (ACT) is a mindfulness-based therapy that focuses on enabling individuals to accept what is out of their control, and to commit to valued actions that enrich their lives. ACT was developed in 1986 by Stephen C. Hayes who began to examine how language and thought influence internal experiences. By emphasizing acceptance instead of avoidance, ACT differs from many other forms of cognitive behavioral therapy. Although not originally designed for CP, ACT has been shown to be efficacious in terms of clinical outcomes, adherence to treatment, and retention, earning the status of a "well-established" treatment for CP from the American Psychological Association. ACT aims to increase psychological flexibility, and has been associated with improved health outcomes in many randomized controlled clinical trials, including three systematic reviews specific to CP. Psychological flexibility is defined as an individual's ability to "recognize and adapt to various situational demands; shift mindsets or behavioral repertoires when these strategies compromise personal or social functioning; maintain balance among important life domains; and be aware, open, and committed to behaviors that are congruent with deeply held values." ACT is a "third wave" behavioral treatment that has been shown to be efficacious for treating CP, as well as co-morbid conditions and factors (e.g., goal selection) related to long-term functional improvement. Additionally, patients who participate in ACT report greater long-term satisfaction compared to CBT. ACT is transdiagnostic and associated with improvements in physical functioning and pain-related disability, as well as decreases in emotional distress regardless of perceived pain intensity.

Resting-state functional magnetic resonance imaging (rsfMRI) allows for data to be collected while individuals with CP rest in the MRI scanner for a short period of time (<10 minutes). Thus, data provides information about the natural state of brain function in CP without having to apply any external sensory or cognitive stimulation. Analysis methods of rsfMRI have focused on multiple regions in the brain, targeting inherent and altered measures of connectivity between brain regions and within brain networks. Further, alterations in brain structure and function have been demonstrated in multiple CP syndromes. Prior imaging research has suggested that CP results in abnormal hyper-connectivity of brain networks associated with self-reflection (default mode, DMN), emotion (salience, SN), and cognitive control (frontal parietal, FPN) networks. While ACT has been successful in helping those with CP create a more functional and personally meaningful life, a critical gap in the understanding of the neural mechanisms underlying ACT remains.

Only two prior investigations have used fMRI to assess neural mechanisms of ACT-based interventions for CP. The first investigated task fMRI activation using pressure evoked pain. Participants with fibromyalgia showed increased activation in the ventrolateral prefrontal cortex (vlPFC) and orbitofrontal cortex (OFC) post-ACT after 12 weeks of ACT. Additionally, results showed pain-evoked changes in connectivity between the vlPFC and thalamus after ACT. Researchers in the second investigation conducted an 8-week ACT intervention vs. health education control (HEC) for participants with comorbid CP and opioid addiction. Focusing on DMN and pain regions in the brain, participants receiving ACT exhibited decreased activation during evoked pain in the middle frontal gyrus (MFG), inferior parietal lobule (IPL), insula, anterior cingulate cortex (aCC), posterior cingulate cortex (pCC), and superior temporal gyrus (STG) compared with HEC participants.

In the present study, ACT was delivered to nine women with CP. fMRI was used to identify changes in brain networks underlying ACT-related behavioral outcomes in CP. Based on prior work examining ACT in CP, the investigators hypothesize that: (1) ACT will reduce connectivity strength within and between the DMN, SN, and FPN, and that (2) changes in connectivity strength will correlate with changes in behavioral outcomes from pre- to post-ACT.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* Chronic musculoskeletal pain duration for greater than or equal to 3 months
* Pain interference greater than or equal to 4 on Brief Pain Inventory (BPI; 0-10 scale)
* No known contraindication to participate
* Access to regular transportation
* No plans to move or become pregnant in the next 3 months
* MRI safe
* Personal cell phone with the ability to receive text messages and access web-based material (e.g. short surveys)

Exclusion Criteria:

* Unstable medical condition, including a movement disorder, such as restless leg syndrome or Parkinson's disease, a neurological disorder such as Alzheimer's disease, history of stroke or brain lesion, a psychiatric disorder such as schizophrenia or bipolar disorder
* Significant cognitive impairment
* Pregnancy(a test must be conducted on each scan day)
* A recent history of: cancer, malignancy, accident or trauma, palliative care, acupuncture, chiropractic care, cognitive-based psychotherapy, other form of alternative care to treat pain condition
* Metal in the body of any sort - implants, pacemaker, pins, screws

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Network Based Statistic (NBS) from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-weeks post-treatment (within 1 week after treatment completion) fMRI scan data
  Derived from fMRI data, the NBS the Network Based Statistic (NBS) is used to examine changes in functional connectivity from pre-to post ACT.

SECONDARY OUTCOMES:
Change in self-reported measures of depression from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-week post-treatment (within 1 week after treatment completion) assessment data
  Depression Scale, as measured by the Center for Epidemiologic Studies Scale (CES-D)
Change in self-reported measures of satisfaction with social role from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-week post-treatment (within 1 week after treatment completion) assessment data
  NIH Toolbox Neuro-QoLTM (Quality of Life in Neurological Disorders) scale

OTHER OUTCOMES:
Change in self-reported measures of pain acceptance from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-week post-treatment (within 1 week after treatment completion) assessment data
  Chronic Pain Acceptance Questionnaire (CPAQ)
Change in self-reported measures of pain interference from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-week post-treatment (within 1 week after treatment completion) assessment data
  NIH Patient-Reported Outcome Measurement Information System (PROMIS) scale
Change in self-reported measures of acceptance and action from pre-to post-ACT | Measured by comparison of pre-treatment (baseline) and 4-week post-treatment (within 1 week after treatment completion) assessment data
  Acceptance & Action Questionnaire (AAQ-II)

CONTACTS AND LOCATIONS:
Locations (1):
- Communication Science and Disorders Research Laboratory, University of New Hampshier, Durham, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vowles KE, McCracken LM, McLeod C, Eccleston C. The Chronic Pain Acceptance Questionnaire: confirmatory factor analysis and identification of patient subgroups. Pain. 2008 Nov 30;140(2):284-291. doi: 10.1016/j.pain.2008.08.012. Epub 2008 Sep 27. PMID 18824301
- [Background] Hemington KS, Wu Q, Kucyi A, Inman RD, Davis KD. Abnormal cross-network functional connectivity in chronic pain and its association with clinical symptoms. Brain Struct Funct. 2016 Nov;221(8):4203-4219. doi: 10.1007/s00429-015-1161-1. Epub 2015 Dec 15. PMID 26669874
- [Background] Napadow V, LaCount L, Park K, As-Sanie S, Clauw DJ, Harris RE. Intrinsic brain connectivity in fibromyalgia is associated with chronic pain intensity. Arthritis Rheum. 2010 Aug;62(8):2545-55. doi: 10.1002/art.27497. PMID 20506181
- [Background] Sporns O. Graph theory methods: applications in brain networks. Dialogues Clin Neurosci. 2018 Jun;20(2):111-121. doi: 10.31887/DCNS.2018.20.2/osporns. PMID 30250388
- [Background] van Ettinger-Veenstra H, Lundberg P, Alfoldi P, Sodermark M, Graven-Nielsen T, Sjors A, Engstrom M, Gerdle B. Chronic widespread pain patients show disrupted cortical connectivity in default mode and salience networks, modulated by pain sensitivity. J Pain Res. 2019 May 29;12:1743-1755. doi: 10.2147/JPR.S189443. eCollection 2019. PMID 31213886
- [Background] Zalesky A, Fornito A, Bullmore ET. Network-based statistic: identifying differences in brain networks. Neuroimage. 2010 Dec;53(4):1197-207. doi: 10.1016/j.neuroimage.2010.06.041. Epub 2010 Jun 25. PMID 20600983
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996